CLINICAL TRIAL: NCT04086212
Title: Ultrafiltration Efficacy of a PD Solution Containing Icodextrin-Xylitol-Carnitine Compared to Icodextrin Alone, an Exploratory Study.
Brief Title: Ultrafiltration Efficacy of a PD Solution Containing Icodextrin-Xylitol-Carnitine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study never started
Sponsor: Iperboreal Pharma Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IP-001-10
Record Dates: First submitted 2019-09-02; First posted 2019-09-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2022-03

CONDITIONS: End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Icodextrin; Xylitol; Peritoneal Dialysis; Dialysis Solutions

STUDY DESIGN:
Intervention Model Description: Randomized cross-over, controlled, open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IXC Peritoneal dialysis solution (Experimental): IXC (Icodextrin, Xylitol and L-Carnitine) Peritoneal dialysis solution
  Interventions: Drug: Icodextrin, xylitol and carnitine solution for peritoneal dialysis
- Icodextrin (Active Comparator): Extraneal® (7.5% Icodextrin) Peritoneal dialysis solution
  Interventions: Drug: EXTRANEAL 7.5G/100Ml Peritoneal Dialysis Solution

INTERVENTIONS:
Drug: Icodextrin, xylitol and carnitine solution for peritoneal dialysis — Patients will receive a long dwell exchange for three days.
  Other Names: IXC
  Arms: IXC Peritoneal dialysis solution
Drug: EXTRANEAL 7.5G/100Ml Peritoneal Dialysis Solution — Patients will receive a long dwell exchange for three days.
  Other Names: icodextrin
  Arms: Icodextrin

SUMMARY:
Randomized, cross-over, controlled, open label study. The aim of this study is to demonstrate that glucose may completely be replaced by a combination of xylitol and carnitine in the bimodal PD solution for long dwell exchange.

DETAILED DESCRIPTION:
The use of a solution icodextrin, xylitol and carnitine (IXC) as the osmotic agent in dialysate for the long dwell exchange provides sustained ultrafiltration (UF) through colloid osmosis, allowing a consistent reduction in extracellular fluid volume without the expected fall in urine output. The other major advantage of IXC is the reduced exposure and absorption of glucose as the main osmotic agent in PD therapy. The aim of this study is to demonstrate that glucose may completely be replaced by a combination of xylitol and carnitine in the bimodal IXC-based PD solution. Compared to glucose, indeed, carnitine and xylitol are extremely stable naturally occurring compounds, even at temperatures higher than those used to steam-sterilize infusional product. As a consequence, xylitol and carnitine may represent better alternatives than glucose as an osmotic ingredient both from the manufacturing and biocompatibility standpoints. Moreover, xylitol and carnitine have an excellent safety profile and possess distinct systemic actions, which are more favorable than glucose.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of ESRD and have been on Continuous Ambulatory Peritoneal Dialysis (CAPD) or Automated Peritoneal Dialysis (APD) for at least 3 months
* A stable clinical condition during the two weeks immediately prior to randomization
* Blood hemoglobin concentration above 8,5 g/100ml
* Has not experienced peritonitis episodes in the last 3 months
* Treated with Extraneal for at least 1 month
* Peritoneal Equilibration Test (PET) performed in the last three months
* Has understood and signed the Informed Consent Form.

Exclusion Criteria:

* History of drug or alcohol abuse in the six months prior to entering the protocol
* Acute infectious condition
* History of severe congestive heart failure and clinically significant arrhythmia
* Malignancy within the past 5 years, including lymphoproliferative disorders
* A medical condition that, in the judgment of the Investigator, would jeopardize the patient's safety following exposure to study drug
* A clinically relevant under-hydration as judged by the treating physician
* History of L-Carnitine therapy or use in the month before entering the study
* Received any investigational drug in the 3 months before entering the study
* Pregnancy, lactation, fertility age without protection against pregnancy by adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Net-ultrafiltration | Changes from baseline value at the end of each product administration period (3 days)
  Net Ultrafiltration at 10 hours (duration of long dwell), in mL, is defined as the difference between the weight of drained volume and weight of the effluent (fill volume).

SECONDARY OUTCOMES:
Sodium removal | Calculated every day for 3 days during each product administration period.
  Net sodium removal will be calculated as the difference between the total amount of sodium drained at end of long dwell (10 hours) and its measure value in the dialysate at time 0 before the initial infusion. Sodium will determined by the hospital laboratory.
Carnitine plasmatic level | Every day for 3 days during each product administration and during the wash-out period
  Carnitine plasmatic level is assessed by chemical analysis of patient's plasma samples.
Xylitol plasmatic level | Every day for 3 days during each product administration and during the wash-out period.
  Xylitol plasmatic leve is assessed by chemical analysis of patient's plasma samples.
Xylitol absorption | Every day for 3 days during each product administration
  Xilitol absorption is determined by calculating the difference (in grams) between the amount of xylitol (measured by lab analysis) in plasma and the amount of xylitol in the patient's dialysis solution administered.
Adverse Events | Through study completion, an average of 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Bonomini, MD, Principal Investigator — Institute of Nephrology, University of Chieti, Italy

IPD SHARING:
Plan to Share IPD: No